CLINICAL TRIAL: NCT03284632
Title: e-Cigarettes: Formaldehyde DNA Adducts, Oxidative Damage, and Potential Toxicity and Carcinogenesis
Brief Title: e-Cigarette - DNA Adducts
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017NTLS040
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Smoking; Cigarette Smoking; Electronic Cigarettes
Keywords: Tobacco; E-Cigarettes; Toxicants; Formaldehyde DNA Adducts; Oxidative Damage
MeSH Terms: conditions — Smoking; Cigarette Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy Coat, Serum, Plasma, Urine, Buccal Cells, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers
- E-cigarette users
- Non-smokers

SUMMARY:
This study will examine the level of toxicity of e-cigarette use compared to smokers and nonsmokers including inflammation markers, toxicant and carcinogen exposure. Additionally, the study will look at the effect of varying voltage levels for e-cigarette users.

DETAILED DESCRIPTION:
In this observational study, e-cigarette users, smokers, and non-users of e-cigarette or tobacco products (up to 134 per group) will be recruited from the Minneapolis-St. Paul area. This research will be conducted at the Tobacco Research Programs at the University of Minnesota. Subjects are screened for eligibility over the phone. If eligible after the phone screen, participants will be invited to attend orientation screening visit in the clinic where consent will be obtained and subjects will complete forms about their tobacco and e-cigarette use and medical history. Subjects who eligible will be asked to return for six visits over the course of six months.

At these appointments, subjects will provide biological specimen samples (buccal cells, urine and blood). Saliva will be collected before and after a smoking or vaping session. Non-users will only have 1 saliva collection.

Subjects will be asked for information pertaining to and e-cigarette and tobacco use and overall health.

ELIGIBILITY:
Inclusion Criteria:

* Good physical health with no unstable medical conditions; Able to provide written informed consent; Stable and good mental health;

Meet criteria for 1 of three groups:

1. Regular smokers confirmed by CO;
2. E-cigarette users (exclusive e-cigarette use for 3 months); Non-Tobacco Users
3. Non-smokers

Exclusion Criteria:

* Unstable medical condition Not willing to attend visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited locally within reasonable distance from the University of Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
DNA Adducts | 6 months
  Formation of Formaldehyde DNA Adducts in oral cells before and after smoking or vaping

SECONDARY OUTCOMES:
Urinary 8-iso-PGF-2α | 6 months
  Stability of Urinary 8-iso-PGF-2α (biomarkers of oxidative damage) over a 6-month sample period
Urinary PGEM | 6 months
  Stability of Urinary PGEM (biomarker of inflammation) over a 6-month sample period
C-reactive protein | 6 months
  Stability of C-reactive protein in serum (biomarker of inflammation) over a 6-month sample period
TNE | 6 months
  Total Nicotine Equivalents (nicotine exposure) over a 6-month sample period

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hecht, Phd, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States